CLINICAL TRIAL: NCT04724447
Title: EXPERIMENTAL ANTIVIRAL TREATMENT OF CYTOMEGALOVIRUS IN DEPRESSION: AFFECTIVE, NEURAL, AND INFLAMMATORY MECHANISMS
Brief Title: ANTIVIRAL TREATMENT OF CYTOMEGALOVIRUS IN DEPRESSION
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Laureate Institute for Brain Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-001
Record Dates: First submitted 2021-01-22; First posted 2021-01-26 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Valganciclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valganciclovir (Experimental): 900 milligrams (mg) valganciclovir (VGCV) to be taken orally once per day for 8 weeks.
  Interventions: Drug: Valganciclovir
- Placebo (Placebo Comparator): Placebo equivalent of 900 milligrams (mg) VGCV to be taken orally once per day for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valganciclovir — 2 x 450mg VGCV tablets
  Arms: Valganciclovir
Drug: Placebo — Placebo equivalent of 900mg/day VGCV
  Arms: Placebo

SUMMARY:
This study aims to determine whether treatment of CMV positive (CMV+) individuals with major depressive disorder (MDD) with valganciclovir (VGCV) alters neural circuitry, reduces inflammation, and improves depressive behavior and symptoms to a greater extent than placebo. In this double-blind, randomized placebo-controlled, parallel group trial, 24 individuals with a Quick Inventory of Depressive Symptomatology-Self Report (QIDS-SR) scale score ≥ 14 will be enrolled to participate in an 8-week treatment study. Participants will be randomized with a 1-1 ratio to receive 900 milligrams (mg) VGCV or placebo to be taken orally once per day. Participants will complete a 2-hour pre-screen, a baseline blood-draw, clinical evaluation, and MRI scan (visit 2), a clinical evaluation, blood draw, and MRI scan at week 4 (visit 6), and a clinical evaluation, blood draw, and MRI scan at week 8 (visit 10). Weekly telephonic visits to assess depressive symptoms and side effects will held between the in-person assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-65 years
4. Diagnosis with major depressive disorder (MDD)
5. Current symptoms of depression, that is, a QIDS-SR score ≥14.
6. Unmedicated for at least 4 weeks (8 weeks for fluoxetine).
7. In good general health as evidenced by medical history, physical exam, and safety labs
8. Ability to take oral medication and be willing to adhere to the VGCV regimen
9. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional 4 weeks after the end of VGCV administration
10. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during the study and for at least 90 days after the study.
11. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

    Exclusion Criteria:

    General Exclusion Criteria:
    * Pregnancy
    * Breast-feeding
    * Unwillingness to avoid pregnancy during the study due to the possible teratogenic effects of valganciclovir

    Medical Conditions:
    * Moderate to severe traumatic brain injury (>30 min. loss of consciousness or >24 hours posttraumatic amnesia) or other neurocognitive disorder with evidence of neurological deficits.
    * Presence of co-morbid medical conditions not limited to but including cardiovascular (e.g., history of acute coronary event, stroke) and neurological diseases (e.g., Parkinson's disease), as well as pain disorders.
    * Presence of co-morbid inflammatory disorders such as rheumatoid arthritis or other autoimmune disorders.
    * Presence of an uncontrolled medical condition that is deemed by the investigators to interfere with the proposed study procedures, or to put the study participant at undue risk.
    * Presence of a chronic infection (e.g. HIV) that may elevate pro-inflammatory cytokines.
    * Presence of an acute infectious illness (e.g. SARS CoV-2) or receipt of a vaccination in the week prior to enrollment.

    Psychiatric Disorders:
    * Current significant suicidal ideation (intent to commit suicide or making specific plans for suicide)
    * Suicide attempt within the last 6 months
    * Lifetime history of schizophrenia, schizophreniform, schizoaffective disorder, delusional disorder
    * History of a manic or hypomanic episode not better accounted for by substance use
    * Moderate to severe substance use disorder within the last year, excluding cannabis or nicotine use disorder
    * Moderate or severe alcohol use disorder
    * Positive urine toxicology (except cannabis)

    Contraindications to Valganciclovir:
    * Myelosuppressive chemotherapy or radiation therapy
    * Absolute neutrophil count < 500/mm3
    * Platelet count < 25,000/mm3
    * Hemoglobin < 8g/dL
    * Impaired renal function (estimated glomerular filtration rate <60mL/minute/1.73m2)
    * Sensitivity to VGCV, ganciclovir or other nucleoside analogues
    * Medications that could interact with VGCV (see below):

    Prohibited Medications Abacavir Lamivudine, 3TC Amikacin Aminoglycosides Amphotericin B cholesteryl sulfate complex (ABCD) Amphotericin B lipid complex (ABLC) Amphotericin B liposomal (LAmB) Amphotericin B Aprotinin Bacitracin Bictegravir; Emtricitabine; Tenofovir Alafenamide Cisplatin Colchicine; Probenecid Cyclosporine Dapsone Darunavir; Cobicistat; Emtricitabine; Tenofovir alafenamide

    Didanosine, ddI:

    Doravirine; Lamivudine; Tenofovir disoproxil fumarate Doxorubicin Efavirenz; Emtricitabine; Tenofovir Efavirenz; Lamivudine; Tenofovir Disoproxil Fumarate Elvitegravir; Cobicistat; Emtricitabine; Tenofovir Alafenamide Elvitegravir; Cobicistat; Emtricitabine; Tenofovir Disoproxil Fumarate Emtricitabine Emtricitabine; Rilpivirine; Tenofovir alafenamide Emtricitabine; Rilpivirine; Tenofovir disoproxil fumarate Emtricitabine; Tenofovir alafenamide Emtricitabine; Tenofovir disoproxil fumarate Entecavir Flucytosine Gentamicin Hyaluronidase, Recombinant; Immune Globulin Hydroxyurea Imipenem; Cilastatin Immune Globulin IV, IVIG, IGIV Kanamycin Lamivudine; Tenofovir Disoproxil Fumarate Mycophenolate Paromomycin Pentamidine Plazomicin Polymyxin B Streptomycin Sulfamethoxazole; Trimethoprim, SMX-TMP, Cotrimoxazole Tacrolimus Talimogene Laherparepvec Telbivudine Tenofovir Alafenamide Tenofovir, PMPA Tobramycin Trimethoprim Vancomycin Vinblastine Vinca alkaloids Vincristine Liposomal Vincristine Vinorelbine Zidovudine

    Other Medications:
    * Current and/or past regular use of hormone-containing medications (excluding contraceptives)
    * Current use of non-steroid anti-inflammatory drugs that is deemed by the investigators to potentially confound the results of the study or the increase risk of renal impairment (e.g. more than 3 days/week).
    * Current and/or past regular use of immune modifying drugs that target specific immune responses such as TNF antagonists
    * Chronic use of antibiotics such as isotretinoin or minocycline because of their potential effects on the microbiome and immune function.
    * Current and/or past regular use of antiarrhythmic, anti-anginal, and anticoagulant drugs (does not apply where medications are taken for different purpose).
    * Inclusion of individuals reporting other types of medications or supplements not listed or considered thus far will be at the discretion of the PI based on their potential to affect immune function, brain function or brain blood flow.

    Contraindications to MRI:
    * Cardiac pacemaker, metal fragments in eyes/skin/body (shrapnel), aortic/aneurysm clips, prosthesis, by-pass surgery/coronary artery clips, hearing aid, heart valve replacement, shunt (ventricular or spinal), electrodes, metal plates/pins/screws/wires, or neuro/bio-stimulators (TENS unit), persons who have ever been a professional metal worker/welder, history of eye surgery/eyes washed out because of metal, vision problems uncorrectable with lenses, inability to lie still on one's back for 60 minutes; prior neurosurgery; tattoos or cosmetic makeup with metal dyes, unwillingness to remove body piercings, and pregnancy.
    * Claustrophobia severe enough to prevent scanning

    Health Factors:
    * BMI > 38 because of the effects of obesity on pro-inflammatory cytokine activity
    * Clinically significant abnormalities on screening laboratory tests

    Non-English speaking participants:

    • The majority of the assessments proposed for this study have not been translated from English, thus, non-English speaking volunteers will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
White matter integrity of the inferior fronto-occipital fasciculus (IFOF) | 8 weeks
  Mean fractional anisotropy of the IFOF measured with diffusion tensor imaging

SECONDARY OUTCOMES:
Volume of the medial temporal gyrus (MTG) | 8 weeks
  Mean gray matter volume of the MTG measured with structural MRI

OTHER OUTCOMES:
Volume of the orbitofrontal cortex (OFC) | 8 weeks
  Mean gray matter volume of the OFC measured with structural MRI
Inflammatory mediators | 8 weeks
  Serum concentration of inflammatory mediators: CXCL10, sCD14, and TNF measured with ELISA or the Mesoscale Discovery Platform
CD8+ cells | 8 weeks
  Percentage of terminally differentiated CD8+ cells (TEMRA cells) measured with flow cytometry
Anhedonia | 8 weeks
  Symptoms of anhedonia measured with the Snaith-Hamilton Pleasure Scale (SHAPS). Higher scores are indicative of greater anhedonia.
Depression | 8 weeks
  Symptoms of depression measured with the Montgomery-Asberg Depression Rating Scale (MADRS). Higher scores are indicative of more severe depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Laureate Institute for Brain Research, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No